CLINICAL TRIAL: NCT03252275
Title: Use of Simulation Based Education With Peer Learning to Enhance HBB Training for Managing Maternal Newborn and Child Health Emergencies in Rural Uganda: A Cluster-randomized Trial
Brief Title: Peer Learning and HBB in Managing Maternal Newborn and Child Health Emergencies in Rural Uganda
Acronym: SimForLife
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mbarara University of Science and Technology (Other)
Collaborators: University of Calgary (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: MUST 21/06-16
Record Dates: First submitted 2017-08-09; First posted 2017-08-17 (Actual); Last update posted 2017-08-17 (Actual); Status verified 2017-08

CONDITIONS: Maternal, Newborn and Child Health Emergencies

STUDY DESIGN:
Intervention Model Description: We will conduct a parallel comparison of intervention and control arms to measure study endpoints
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Standard HBB and ECEB training with peer learning
  Interventions: Other: Peer learning
- Control (No Intervention): Standard HBB and ECEB training only

INTERVENTIONS:
Other: Peer learning — Peer learning plus HBB and ECEB
  Arms: Intervention

SUMMARY:
The aim of this study is to test an intervention that has potential to improve acute care skills and confidence related to safe delivery and newborn care for mid-level health providers in Uganda by the development of a 'mobile' simulation package including scale-up materials based upon research evidence. In this randomized study investigators will compare the impact of a peer learning package on skills, knowledge and team work regarding newborn care among health workers in rural south western Uganda.

DETAILED DESCRIPTION:
The aim of this study is to test an intervention that has potential to improve acute care skills and confidence related to safe delivery and newborn care for mid-level health providers in Uganda by the development of a 'mobile' simulation package including scale-up materials based upon research evidence. In this randomized study investigators will compare the impact of a peer learning package on skills, knowledge and team work regarding newborn care among health workers in rural south western Uganda.

The cluster randomized study will have two arms; intervention arm receives peer learning program. In this program, two health workers at the same health facility teach each other using case scenarios. The case scenarios will be based on common neonatal conditions such as neonatal sepsis, hypothermia and prematurity.

The two study arms will both receive training on HBB and Essential care for every baby (ECEB)

ELIGIBILITY:
Inclusion Criteria:

* Health workers involved in performing deliveries of mothers at health center IVs and IIIs (i.e, county and subcounty level)

Exclusion Criteria:

* Health facilities based in municipalities, urban dwellings

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 77 (Estimated)
Dates: Start 2017-08-30 (Estimated); Primary Completion 2020-01 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Skills on key maternal, newborn and child health emergency procedures | Change in skills scores at 6 and 12 months from Baseline
  Ability to perform key maternal, new born and child health emergency procedures measured using Multiple choice questions (MCQs). A composite score with a maximum of 100% will be computed from these MCQs

SECONDARY OUTCOMES:
Clinical teamwork scores | Change in CTS scores at 6 and 12 months from Baseline
  Ability to work as a team through communication, sharing roles and completing tasks together measured using the Clinical Teamwork scale (CTS). A composite score will be computed by adding up all the items on the CTS scale. CTS has 15 items, each item with a maximum score of 10

CONTACTS AND LOCATIONS:
Overall Officials: Santorini Data, MD, Principal Investigator — Mbarara University of Science and Technology

IPD SHARING:
Plan to Share IPD: Undecided
Authorization to share data will be sought

REFERENCES:
- [Derived] Data S, Mirette D, Cherop M, Bajunirwe F, Kyakwera C, Robinson T, Josephine NN, Abesiga L, Namata T, Brenner JL, Singhal N, Twine M, Wishart I, McIntosh H, Cheng A. Peer Learning and Mentorship for Neonatal Management Skills: A Cluster-Randomized Trial. Pediatrics. 2022 Aug 1;150(2):e2021054471. doi: 10.1542/peds.2021-054471. PMID 35794462